CLINICAL TRIAL: NCT01975766
Title: A Phase I Trial of a Ketogenic Diet With Concurrent Chemoradiation for Head and Neck Cancer
Brief Title: Ketogenic Diet Phase 1 for Head & Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Bryan Allen (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Nutricia North America (Industry); Holden Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Bryan Allen, Assistant Professor, Department of Radiation Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201309759; 3P30CA086862 (NIH)
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Head and Neck Neoplasms
Keywords: Carcinoma, squamous cell of head and neck; Head and neck cancer; ketogenic diet; radiotherapy; cisplatin
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Diet, Ketogenic; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic diet (Experimental): Ketogenic diet designed to sustain ketone levels through treatment.
  Interventions: Dietary Supplement: Ketogenic diet; Device: External beam radiation therapy

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — A ketogenic diet matching the fat to carbohydrate + proteins in Keto-Cal(R) 4:1 by Nutricia North America.
Device: External beam radiation therapy
  Other Names: radiation therapy; intensity modulated radiation therapy; IMRT

SUMMARY:
This study investigates if using a very low carbohydrate diet during combined chemotherapy and radiation therapy is safe and if it can be tolerated by patients.

DETAILED DESCRIPTION:
Standard treatment for head & neck cancer often includes chemotherapy concurrent with radiation therapy (chemoradiation).

This study is a phase I trial to determine the safety of dietary manipulation during chemoradiation for head & neck cancer. Specifically, pre-clinical data from mouse studies indicates a ketogenic diet increases tumor cell killing.

Participants will:

* Utilize a specialized ketogenic diet designed by bionutritional services of the clinical research unit. This diet begins 2 days before chemoradiation and continues through at least 5 weeks of chemoradiation.
* Have blood drawn for research purposes weekly to determine measurements of oxidative stress
* Have urine collected sporadically through the study to determine measurements of oxidative stress
* Keep a diary of concomitant medications, side effects, and blood sugars
* Have follow-up to monitor for outcomes and overall survival

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented squamous cell carcinoma of the oropharynx, larynx or hypopharynx. HPV status will not be assessed for eligibility; while HPV status may affect response to therapy, efficacy is not an outcome measure for this phase I study.
* Candidate for primary chemoradiation as decided by an interdisciplinary team including otolaryngology, medical oncology, and radiation oncology.
* Cancer should be staged via AJCC as stage II, III or IVa.
* Age ≥ 18 years
* ECOG performance status 0-2 (Karnofsky > 50%, see Appendix A).
* Patients must have normal organ and marrow function as defined below:
* leukocytes ≥ 3,000/mm3
* absolute neutrophil count ≥ 1,500/mm3
* platelets ≥ 100,000/mm3
* total bilirubin < 1.5 mg/dl
* Hgb A1C < 8%
* AST(SGOT) < 2 X institutional upper limit of normal
* creatinine < 1.5 X institutional upper limit of normal OR calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Not pregnant. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Life expectancy of 3 or less months.
* Prior neck and/or upper thoracic radiotherapy that would cause an overlap of treatment fields.
* Prior therapy to the head and neck, with the intent to treat, the current diagnosis of head & neck cancer.
* Known / established G6PD (glucose-6-phosphate dehydrogenase) deficiency.
* Chronic system corticosteroids for any reason (inhaled corticosteroids are allowed). Pre-medication for chemotherapy is acceptable.
* Other investigational agents/therapy with the intention to treat the disease under study (observational or imaging trials are acceptable).
* Uncontrolled diabetes defined as a hemoglobin A1C level > 8% (therapeutic action is indicated at greater than 8%).
* Diabetes is not exclusionary provided the patient is not maintained with either oral medications or insulin.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements as determined by study team members.
* Pregnant or lactating women: The risks of radiation and chemotherapy to a fetus are well documented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (safety) | weekly for 5 weeks
  Categorize and quantify adverse events in subjects implementing a ketogenic diet while undergoing definitive chemoradiation therapy.

SECONDARY OUTCOMES:
Ketone levels | Daily during treatment for 5 weeks
  Quantify blood ketone levels via both finger-stick prior to daily radiation therapy and weekly lab analysis while on a ketogenic diet. Radiation is administered Monday through Friday only.
Blood glucose levels | daily during treatment for 5 weeks
  Quantify blood glucose levels via finger-stick prior to daily radiation therapy while on a ketogenic diet. Radiation therapy is administered Monday through Friday only.
Oxidative stress parameters | Weeks 1, 2, 3, 4, and 5 of treatment and at 1 month follow-up
  Determine oxidative stress parameters in plasma and urine samples during the course of treatment.
Progression Free Survival (months) | Every 12 months for 60 months
  From date of treatment until the first date of documented progression or date of death, whichever comes first, assessed no less than every 12 months for the first 60 months post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bryan G. Allen, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on clinicaltrials.gov

REFERENCES:
- [Result] Allen BG, Bhatia SK, Buatti JM, Brandt KE, Lindholm KE, Button AM, Szweda LI, Smith BJ, Spitz DR, Fath MA. Ketogenic diets enhance oxidative stress and radio-chemo-therapy responses in lung cancer xenografts. Clin Cancer Res. 2013 Jul 15;19(14):3905-13. doi: 10.1158/1078-0432.CCR-12-0287. Epub 2013 Jun 6. PMID 23743570